CLINICAL TRIAL: NCT06331117
Title: The Impact of Ras/MAPK Pathway Hyperactivation on Bioenergetic Metabolism and Its Effect on Growth Profile and Bone Metabolism
Brief Title: Effect of RAS/MAPK Pathway Hyperactivation on Growth' and Bone' Profile of the RASopathies
Acronym: 3776
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Leoni Chiara, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3776
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: RASopathy; Costello Syndrome; Noonan Syndrome; Cardio-Facio-Cutaneous Syndrome
MeSH Terms: conditions — Costello Syndrome; Noonan Syndrome; Cardiofaciocutaneous syndrome | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): Multiomics profiling of the RASopathies
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — Multiomics profiling

SUMMARY:
Costello syndrome (CS) and cardio-facio cutaneous syndrome (CFCS) belongs to RASopathies, a group of multisystemic disorders caused by unregulated signalling through the RAS/MAPK pathway, an intracellular signalling pathway regulating multiple processes such as cellular proliferation, differentiation, survival, apoptosis and also contributing to oncogenesis. They share a recognizable facial appearance, aged appearance, growth delay, muscle-skeletal anomalies, heart defects, neuropsychological features, skin and ocular abnormalities, and cancer predisposition.

Even though life expectancy of individuals with CS and CFCS has increased in the last years due to the improvement of patients' care and a more effective prevention of comorbidities, some of the most challenging aspects impacting on everyday living such as growth failure, accelerate senescence and skeletal-muscle defects, still need to be fully understood. This statement underlies the need to improve clinical research protocols with more innovative techniques (multi-omics profiling) in order to better understand the effect of RAS/MAPK pathway hyperactivations on different systems and to define possible personalized treatments.

DETAILED DESCRIPTION:
Multiomics profiling of the RASopathies

ELIGIBILITY:
Inclusion Criteria:

* Clinical and molecularly confirmed diagnosis of a RASopathy

Exclusion Criteria:

* Only clinical diagnosis of a RASoapthy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Metabolomic profile of the RASopathies | 3 years
  To perform metabolomic profile in all enrolled RASopahty patients

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Leoni, MD, PhD, Principal Investigator — Fondazione Policlinico A. Gemelli, IRCCS
Locations (1):
- Department of Woman and Child Health and Public Health, Fondazione Policlinico A. Gemelli, IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No